CLINICAL TRIAL: NCT06585501
Title: Treatment and Testing Patterns in HER2-positive Unresectable and Advanced Gastric/ Gastroesophageal Junction Cancer in China: A Retrospective Real-world Study (REHEARSAL)
Brief Title: A Study of Treatment Patterns in HER2-positive Unresectable and Advanced Gastric/ Gastroesophageal Junction Cancer in China
Acronym: REHEARSAL
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: DS8201-0014-NIS-MA
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Cancer
Keywords: Gastric Cancer; Gastroesophageal Junction Cancer; HER2; Real-world
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GC/GEJC: Patients diagnosed with locally advanced unresectable or metastatic HER2-positive GC/GEJC
  Interventions: Other: No drug

INTERVENTIONS:
Other: No drug — This is a non-interventional study and no study drug will be provided.

SUMMARY:
This study will be conducted to retrospectively evaluate the treatment patterns in first-line, second-line, and subsequent lines of therapy for HER2-positive Gastric Cancer/Gastroesophageal Junction Cancer (GC/GEJC) patients.

DETAILED DESCRIPTION:
This is a multicenter, non-interventional, retrospective real-world study to analyze the treatment patterns for patients with GC/GEJC in the first-line, second-line, and subsequent lines of treatment. The study will also assess different HER2 sample types, testing methods, and HER2 re-biopsy situations. By evaluating the treatment and testing patterns in clinical practice, this study aims to provide evidence and recommendations for improving the strategies for the treatment and testing of HER2-positive GC/GEJC patients.

ELIGIBILITY:
Inclusion criteria

* Patients with pathologically diagnosed locally advanced unresectable or metastatic GC/GEJC (limited to those diagnosed since October 1, 2017) and initiating first-line treatment between January 1, 2018, and March 31, 2023
* Patients aged ≥ 18 years at the time of diagnosis with locally advanced unresectable or metastatic GC/GEJC; HER2-positive status2, determined by either tissue samples from the first biopsy or liquid biopsy samples (if a patient has both tissue and liquid biopsy samples, tissue samples will be the standard).

Exclusion criteria

* Patients with other primary malignant tumors
* Patients enrolled in clinical trials and receiving active anti-cancer therapy after July.1, 2017 (excluding retrospective studies).
* Patients with critical missing data in medical records or otherwise deemed for inclusion by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with locally advanced unresectable or metastatic HER2-positive GC/GEJC after October 1, 2017, and initiating first-line therapy between January 1, 2018, and March 31, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 805 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients receiving first-line, second-line, and third-line anti-tumor regimens | 72 months

SECONDARY OUTCOMES:
Percentage of HER2 sample type and testing method among patients with a first diagnosis of locally advanced or metastatic HER2-positive GC/GEJC | 72 months
Percentage of re-biopsies and re-biopsies with HER2-positive results among patients with a first diagnosis of locally advanced or metastatic HER2-positive GC/GEJC | 72 months
Real-world Progression-Free Survival | 72 months
Real-world Time to Discontinuation | 72 months
Real-world Time to Next Treatment 1 | 78 months
Overall Survival | 78 months

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Beijing Cancer Hospital, Beijing
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Affiliated Cancer Hospital of Shandong First Medical University, Jinan
  - Liaoning Cancer Hospital & Institute, Shenyang
  - The First Hospital of China Medical University, Shenyang
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan

IPD SHARING:
Plan to Share IPD: No